CLINICAL TRIAL: NCT06341504
Title: Messages de prévention Sur Les Appareils de Loterie vidéo : Effets Sur Les Comportements et Les Cognitions [Prevention Messages for Electronic Gambling Machines: Effects on Behaviours and Cognitions]
Brief Title: Prevention Messages for EGMs: Effects on Behaviours and Cognitions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benjamin Galipeau (Other)
Collaborators: Fonds de recherche du Québec - Société et culture (Unknown); Fonds pour la prévention et le traitement du jeu (Unknown)
Responsible Party: Sponsor-Investigator, Benjamin Galipeau, Ph.D. candidate, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ALVMsg2023; 263472 (Other Grant/Funding Number: Fonds de recherche du Québec - Société et culture)
Record Dates: First submitted 2024-02-14; First posted 2024-04-02 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Gambling
Keywords: Prevention messages; Pop-up messages; Prevention; Gambling; Harmful gambling; Responsible gambling; Harm reduction; Communication; Self appraisal
MeSH Terms: conditions — Gambling; Harm Reduction; Communication

STUDY DESIGN:
Intervention Model Description: Stratified block randomization assignment. Blocks are size 4 and strata are divided on problem gambling severity using PGSI categories. Two conditions:
  * Experimental: Regular gambling session + Prevention pop-up messages
  * Active Comparator: Regular gambling session
  Three assessment phases:
  * Pre-experiment. Telephone interview before the gambling session. Measures baseline characteristics and schedule the gambling session. Usually done within a couple of days following an application to participate.
  * Experiment. Gambling session in the laboratory. Behaviour is continuously measured starting with the first time the participant puts money in the EGM to participant choosing to end their gambling session. Duration is limited to 2 hrs (unbeknownst to participant). Session is scheduled days to weeks after the Pre-experiment, depending on participant's availability.
  * Post-experiment. Debriefing and post-experiment interview. Done right after the gambling session is ended.
Who Masked: Participant
Masking Description: Participants are recruited under the false pretense of evaluating the realism of a gambling session in a laboratory replicating a bar environment. While the participants in the experimental group should notice the novel prevention messages, before debriefing, for all they know, there are no groups to be assigned to. Therefore they would not be aware, that there are two different groups, nor that this study tests the effects of prevention pop-up messages.
  Note that masking becomes "open label" after debriefing. Indeed, after being informed of the true goals of this study, participants will easily be able to determine in which group they were assigned based on what occured during their gambling session. Though, gambling behaviours are recorded before debriefing and won't be affected by unmasking.
  There is no functional way to mask group assignment to the members of the research team. However, the randomization procedure assures that allocation is purely random.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention pop-up messages (Experimental): Same as active comparator with the addition of prevention pop-up messages delivered during the gambling session on a fixed presentation schedule.
  Due to hardware limitations on the EGMs' part, the prevention messages presented only alter what is shown on the play screen (they fill it completely, hiding the game), but can't pause the game per se. The EGMs' buttons, sound, and music are still operational while the message is shown. While disrupting play flow, this still lets the participant place bets (albeit without seeing what is going on).
  Interventions: Behavioral: Prevention pop-up messages; Behavioral: Mandatory time limit; Behavioral: Responsible gambling information; Device: Electronic gambling machine (model IGT GL20); Device: Square terminal
- Regular gambling session control (Active Comparator): Gambling session on EGMs in a room replicating a bar (subdued light, music, bar paraphernalia, fake liquor on display, research assistant acting as barman and selling non-alcoholic soft drinks and chips).
  Participants are invited to participate under the false pretense of giving their opinion on the realism of the bar replica and overall feeling of the gambling session in it. They are told that: (a) they are free to gamble as much and for as long as they like; (b) they are allowed to take breaks; (c) gambling is to be done with their own money; (d) the only compensation for participation are winnings that could be made while gambling; (e) net winnings across their whole session are paid up to $500, but losses are real. Lost money is given back after debriefing (see Study Detailed Description).
  Interventions: Behavioral: Mandatory time limit; Behavioral: Responsible gambling information; Device: Electronic gambling machine (model IGT GL20); Device: Square terminal

INTERVENTIONS:
Behavioral: Prevention pop-up messages — Messages are shown full screen on the EGM's play screen on a fixed presentation schedule. Clock of the gambling session starts the first time the participant puts money in the EGM. From this event, messages are shown at those timepoints: [1] +10 minutes; [2] +40 minutes; [3] +70 minutes; [4] +100 minutes. Messages block the screen for 15 seconds before automatically closing. Up to 4 different messages are presented during the gambling session. Order is determined by sortition without replacement.
  Messages have a warning heading "Caution!". Content is, from top to bottom: (a) time spent gambling from beginning; (b) warning that gambling could lead to serious monetary loss; (c) 1 of 4 self-appraisal phrases about current gambling behaviour; (d) advice to the participant that a break could help choose what is best for them; (e) countdown before the message closes itself; (f) Health department logo is shown in the lower right corner as a more "neutral" endorsement of the messages.
  Arms: Prevention pop-up messages
Behavioral: Mandatory time limit — Activated either when (a) the previous time limit is up; or (b) the player bank meter reaches $0. When the previous time limit is up, a pop-up takes up the upper third of the play screen and requires the player to set a new time limit using one of five choice buttons (four firsts buttons: 15, 30, 45 or 60 minutes; fifth button: cash out, which prints a receipt and ends the gambling session). As the EGM cannot track who is playing, there are no limits on consecutive gambling sessions. When the player's bank meter reaches $0, the the pop-up described above appears as soon as new money is inserted in the EGM, no matter if the previous time limit is up or not.
Behavioral: Responsible gambling information — Located in a submenu accessed through a button on the main touch screen. This open a window which contains basic information on randomness and responsible gambling advice. The information is presented in small white font on a black background.
Device: Electronic gambling machine (model IGT GL20) — EGM model currently in use in Quebec, Canada, the location where this study is conducted. The EGMs used in this study are fully functional and unaltered except for the presentation of prevention pop-up messages in the experimental arm of this study. These machines are equipped with basics responsible gambling features, the two main ones described in this section (i.e. "Mandatory time limit"; "Responsible gambling information"). Wins/losses sequence is fully randomized and not determined beforehand.
  Other Names: EGM
Device: Square terminal — This terminal allows for buying non-alcoholic beverages (soft drinks or coffee) and chips during the experimentation. This is done to enhance the realism of the bar setting. It also allows for real cash withdrawal from bank account during gambling session. Quebec's code of conduct for EGMs commercialization prohibits retailers from having an ATM near their EGMs, and prohibits them from lending money to consumers or withdrawing cash for them to gamble. However, this rule is not always followed in practice. For this study, participants will be allowed to withdraw from their bank account, at the bar counter, if they ask for it. However, this will not be offered to them upfront.

SUMMARY:
The goals of this randomized controlled trial are to test the manifold effects of prevention pop-up messages on participants' behaviours, cognitions and affects. This study is conducted among regular EGMs' players (defined as having played EGMs at least once every two weeks for the past 12 months) who are not classified as probable pathological gamblers by the PGSI.

After answering a series of short questionnaires by phone, participants are asked to schedule a gambling session which is done in a laboratory on the university's campus. This laboratory replicates a typical bar, and is equipped with real EGMs. Participants are recruited under the false pretense of giving their opinion on the realism of the bar replica, and on the overall feeling of the gambling session in it. They are told that: (a) they are free to gamble as much and for as long as they like; (b) they are allowed to take breaks; (c) gambling is to be done with their own money; (d) the only compensation for participation are the potential winnings made while gambling; (e) net winnings across their whole session are paid, but losses are real. There is only one participant at a time in the laboratory for the gambling session.

After having stopped by their own volition (some exceptions apply, see "Detailed Description" for further details), participants are debriefed on the real goals of this study and reimbursed any incurred losses while gambling. They are then be asked to answer another series of questionnaires.

DETAILED DESCRIPTION:
EGMs and online gambling are the reputedly most damaging gambling type from a public health perspective. Pop-up messages are often used as a responsible gambling (RG) measure to prevent harm for these screen-based types of gambling. Despite some evidence of effectiveness in the literature for these messages, limitations persists, among which low ecological validity is of particular concern.

Indeed, gambling studies set in a controlled environment, usually a laboratory setting, often require participants to engage in a gambling task while wagering some form of virtual credits or money provided upfront by the researchers as a compensation for participation. Their behaviour is then assumed alike what would happen in a real gambling setting, even though gamblers are not risking their own money. Surprisingly, this assumption has not been subject to much scientific scrutiny. Moreover, some studies provide data which seems to contradict this assumption.

This study address this limitation by heightening the realism factor. This study starts with an intake interview by phone to evaluate eligibility, PGSI category, sociodemographic characteristics, gambling behaviours on EGMs (past 12 months), general level of fun while playing EGMs (past 12 months) and perceived self-control while playing EGMs. Participants are then asked to schedule a gambling session which is done in a laboratory on the university's campus. This laboratory replicates a typical bar, and is equipped with real EGMs. Participants are recruited under the false pretense of giving their opinion on the realism of the bar replica, and on the overall feeling of the gambling session in it. They are told that:

* They are free to gamble as much and for as long as they like.
* They are allowed to take breaks.
* Gambling is to be done with their own money.
* The only compensation for participation are the potential winnings made while gambling.
* Net winnings across their whole session are paid , but losses are real.

There is only one participant at a time in the laboratory for the gambling session. While in the bar replica, the participant is joined by a research assistant who plays the role of barmaid/barman. The assistant is there for general realism purposes, operating the cash register (Square terminal), and ensuring the general safety of the session. The bar replica has three EGMs, but only one can be played on and used to show the prevention pop-up messages. The other two EGMs are turned on for ambiance purposes, but have their money collector disabled to prevent participants playing on them or switching between EGMs mid-session. Limiting play to only one EGM also eases the recording of gambling behaviours and proper showing of the prevention messages. Participants are told the two "unusable" EGMs are awaiting to be serviced because of their money collector malfunction.

A second research assistant is located in an adjacent room. They are responsible for (a) recording all gambling behaviours using a computer connected to the EGM; and (b) operating the pop-up messages presentation schedule. A spy camera (disguised as a smoke detector) with a live-feed is used to observe gambling related behaviours that can't be recorded by the EGM's computer (e.g. taking a break).

The gambling session ends when the participant cashes out and unambiguously tell the research assistant they want to end their session. The participant is then brought to an office for a series of questionnaires which are, in order:

* Perception of realism of the bar replica and the gambling session in it.
* Debriefing about the true goals of the study and validation of consent to participate in the study. At this point, participants will be able to guess in which group they were assigned.
* Prevention pop-up messages recall (free and cued recall).
* Cognitive and emotional response to prevention pop-up messages.
* Evaluation of protocol credibility (i.e. if participant really believed they were gambling their own money and were really risking their own money).

Note that while the participant is told they can gamble for as long as they like, in reality there is a 2 hours time limit to the gambling session duration. This time limit is hidden from the participant. The gambling session starts with the first time money is inserted in the EGM by the participant (the "clock" is set at 0 hours) and ends with either the participant ending it of their own volition or upon reaching the time limit (2 hours). Breaks during gambling session are permitted (e.g. for going to the bathroom, for buying snacks from the barman/barmaid, etc.) and don't stop the "clock".

If the participant has not yet ended their gambling session on their own volition upon reaching the 2 hours time limit, they will be asked to take a small break to answer some questions. The existence of a time limit will be communicated to them during the debriefing. In the eventuality of a participant refusing to stop playing or wanting to rapidly quit the laboratory (e.g. because they are angry about losing money), the debriefing will be done earlier, before the questionnaire about their perception of realism of the bar replica and the gambling session in it. While not optimal, early debriefing is nevertheless considered acceptable in order to force the end of the gambling session or to prevent a participant from hastily quitting the study without receiving all the information to make an informed decision about their participation. There will be no more gambling done after debriefing.

Upon debriefing the participant will be reimbursed all money lost (if any).

The mains objectives are to test to what extent do RG pop-up messages affect:

1. Participants' gambling behavior (e.g. money betted, gambling session length, gambling intensity, etc.).
2. Participants' cognitions (e.g. thoughts elicited by messages, perceived effectiveness of message, etc.).
3. Participants' emotions (e.g. enjoyment of gambling, emotional response to messages, etc.).

Secondary objectives are to test:

1. to what extent are the main effects moderated by participants' characteristics (e.g., gender, age, education, PGSI category, etc.).
2. the feasibility of studies conducted in a laboratory setting with the use of real money (or using deception to make the participants believe they are gambling their own money). This objective is answered with four sub-questions:

   * Was it possible to recruit enough participants for the study considering they were confronted with the prospect of loosing their own money by participating in the study and were not guaranteed any compensation other than what they could win on the EGMs?
   * Did the laboratory "bar" replicated well the overall "vibe" of a typical gambling venue with EGMs?
   * Did the participants found their gambling session in the bar replica as realistic as a real one?
   * Did the participants believed they were gambling their own money during the study (i.e. to what extent did the deception worked)?

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old (legal age to gamble in Quebec, Canada, where the study is conducted)
* Functional literacy in french (study is conducted in french and requires reading and understanding simple texts)
* Having played EGMs and least once every two weeks for the past 12 months

Exclusion Criteria:

* Classified as a probable pathological gambler (score ≥ 8 on the PGSI)
* Currently receiving treatment for problem gambling
* Currently under self-exclusion from gambling venues

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants are free to self-identify to their prefered gender. Options are "male", "female" or "other".
Enrollment: 80 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Gambling behaviour (between group) - Gambling session's total duration | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Time elapsed between the first time the participant puts money in the EGM (0h00) to the end of the gambling session. Session's duration is left for the participant to decide. While the participant is told they can play for as long as they like, there is a 2 hrs limit on the session duration. This limit is hidden from the participant. Session's duration includes any breaks taken from gambling on the EGM.
Gambling behaviour (between group) - Total time effectively spent gambling | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Same as Outcome 1 (Gambling session's total duration), but minus breaks taken from gambling on the EGM.
Gambling behaviour (between group) - Number of breaks taken | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Number of breaks taken from gambling on the EGM during the gambling session.
Gambling behaviour (between group) - Mean breaks' duration | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Average duration of breaks' taken from gambling on the EGM over the gambling session's total duration.
Gambling behaviour (between group) - Total breaks duration | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Sum of breaks' duration taken from gambling on the EGM over the gambling session's total duration.
Gambling behaviour (between group) - Mean time elapsed between breaks | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Average time separating any two breaks taken from gambling on the EGM over the gambling session's total duration.
Gambling behaviour (between group) - Money betted (physical) | Assessed at following timepoints from start of gambling session in the laboratory (Experiment phase; 0 hours 0 minutes): [1] +10 minutes; [2] +40 minutes; [3] +70 minutes; [4] +100 minutes; [5] end of gambling session (+2 hours maximum).
  Money physically inserted in the EGM during the gambling session. This is evaluated as a cumulative amount at each timepoint a prevention message is presented in the experimental group and at the timepoint where the participant decides to end their gambling session (max 2h00). Money betted is also evaluated between said timepoints (e.g. between 1h10 and 0h40, between 0h40 and 1h10, etc.).
Gambling behaviour (between group) - Money betted (all) | Assessed at following timepoints from start of gambling session in the laboratory (Experiment phase; 0 hours 0 minutes): [1] +10 minutes; [2] +40 minutes; [3] +70 minutes; [4] +100 minutes; [5] end of gambling session (+2 hours maximum).
  Money betted on the EGM during the gambling session. This is money used to "buy rounds on the EGM", whether it's money physically inserted in the EGM or money won while gambling and betted again.
  This is evaluated as a cumulative amount at each timepoint a prevention message is presented in the experimental group and at the timepoint where the participant decides to end their gambling session (max 2h00). Money betted is also evaluated between said timepoints (e.g. between 1h10 and 0h40, between 0h40 and 1h10, etc.).
Gambling behaviour (between group) - Number of bets placed | Assessed at following timepoints from start of gambling session in the laboratory (Experiment phase; 0 hours 0 minutes): [1] +10 minutes; [2] +40 minutes; [3] +70 minutes; [4] +100 minutes; [5] end of gambling session (+2 hours maximum).
  Number of bets placed on the EGM during the gambling session. This is evaluated as a cumulative number at each timepoint a prevention message is presented in the experimental group and at the timepoint where the participant decides to end their gambling session (max 2h00). Number of bets placed are also evaluated between said (e.g. between 1h10 and 0h40, between 0h40 and 1h10, etc.).
Gambling behaviour (between group) - Gambling speed | Assessed at following timepoints from start of gambling session in the laboratory (Experiment phase; 0 hours 0 minutes): [1] +10 minutes; [2] +40 minutes; [3] +70 minutes; [4] +100 minutes; [5] end of gambling session (+2 hours maximum).
  Number of bets placed on the EGM during the gambling session over a given amount of time (i.e. bets/min).
  This is evaluated at each timepoint a prevention message is presented in the experimental group and at the timepoint where the participant decides to end their gambling session (max 2h00). Gambling speed is also evaluated between said timepoints (e.g. between 1h10 and 0h40, between 0h40 and 1h10, etc.).
Gambling behaviour (between group) - Gambling intensity (physical) | Assessed at following timepoints from start of gambling session in the laboratory (Experiment phase; 0 hours 0 minutes): [1] +10 minutes; [2] +40 minutes; [3] +70 minutes; [4] +100 minutes; [5] end of gambling session (+2 hours maximum).
  Money physically inserted in the EGM during the gambling session over a given amount of time (i.e. $/min).
  This is evaluated at each timepoint a prevention message is presented in the experimental group and at the timepoint where the participant decides to end their gambling session (max 2h00). Gambling intensity is also evaluated between said (e.g. between 1h10 and 0h40, between 0h40 and 1h10, etc.).
Gambling behaviour (between group) - Gambling intensity (all) | Assessed at following timepoints from start of gambling session in the laboratory (Experiment phase; 0 hours 0 minutes): [1] +10 minutes; [2] +40 minutes; [3] +70 minutes; [4] +100 minutes; [5] end of gambling session (+2 hours maximum).
  Money betted on the EGM during the gambling session over a given amount of time (i.e. $/min). This is money used to "buy rounds on the EGM", whether it's money physically inserted in the EGM or money won while gambling and betted again.
  This is evaluated at each timepoint a prevention message is presented in the experimental group and at the timepoint where the participant decides to end their gambling session (max 2h00). Gambling intensity is also evaluated between said timepoints (e.g. between 1h10 and 0h40, between 0h40 and 1h10, etc.).
Perceived self-control while gambling on EGMs (between group) | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Participant's perceived ability to control their gambling behaviour (e.g. sticking to their predetermined limits) over the gambling session's total duration. Evaluated with a 7-points Likert scale (1 = "I never had control" to 7 = "I always had control").
General level of fun while gambling on EGMs (between group) | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Participant's general enjoyment of gambling on EGMS over the gambling session's total duration. Evaluated with a 7-points Likert scale (1 = "I hated it" to 7 = "I loved it").
Psychological reactance to prevention pop-up messages (between group) | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Evaluated based on the Dillard & Shen (2005) method: (a) Induction check (4 items, 7-points Likert scale, 1 = "Strongly disagree, 7 - "Strongly agree"); (b) Anger (4 items, 7-points Likert scale, 1 = "Strongly disagree, 7 - "Strongly agree"); (c) Cognitive response (count of negative thoughts in relation to the pop-up messages); (d) Attitude (7 word pairs, 7-points semantic differential scale).
Perceived behavioural effectiveness of prevention pop-up messages (between group) | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Participant's perceived effectiveness of prevention pop-up messages on modifying their gambling behaviour during the gambling session. Evaluated with two 7-points Likert scale about the perceived effects of the prevention po-up messages on money betted and time spent during the gambling session (1 = "lowered gambling behaviour a lot" to 7 = "heightened gambling behaviour a lot").
Change in gambling behaviours (within group) - Money betted (physical) | Change from Pre-experiment phase (i.e. "intake"; single measurement point; cover past 12 months) at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Money physically inserted in the EGM. Change is evaluated by comparing self-reported betting habits on EGMs for the past 12 months (measured during the pre-experiment phase) and objectively measured money physically inserted in the EGM during the over the laboratory gambling session's total duration (Outcome 8; measured during the experiment phase).
Change in gambling behaviours (within group) - Total time effectively spent gambling | Change from Pre-experiment phase (i.e. "intake"; single measurement point; cover past 12 months) at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Time elapsed between the first time the participant puts money in the EGM to the end of the gambling session.
  Change is evaluated by comparing self-reported typical time spent gambling on EGMs for a single session for the past 12 months (measured during the pre-experiment phase) and objectively measured laboratory gambling session's total duration (Outcome 1; measured during the experiment phase). Note that, unbeknown to the participant, the laboratory gambling session is limited to 2 hrs max.
Change in perceived self-control while gambling on EGMs (within group) | Change from Pre-experiment phase (i.e. "intake"; single measurement point; cover past 12 months) at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Participant's perceived ability to control their gambling behaviour on EGMs (e.g. sticking to their predetermined limits). Evaluated with a 7-points Likert scale (1 = "I never had control" to 7 = "I always had control").
  Change is evaluated by comparing self-reported typical perceived self-control while gambling on EGMs for the past 12 months (measured during the pre-experiment phase) and self-reported perceived self-control while gambling on EGMs over the laboratory gambling session's total duration (Outcome 14; measured in the post-experiment phase).
Change in general level of fun while gambling on EGMs (within group) | Change from Pre-experiment phase (i.e. "intake"; single measurement point; cover past 12 months) at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Participant's general enjoyment of gambling on EGMs. Evaluated with a 7-points Likert scale (1 = "I hated it" to 7 = "I loved it").
  Change is evaluated by comparing self-reported typical level of fun while gambling on EGMs for the past 12 months (measured during the pre-experiment phase) and self-reported level of fun while gambling on EGMs over the laboratory gambling session's total duration (Outcome 15; measured in the post-experiment phase).

SECONDARY OUTCOMES:
Perceived realism - Gambling location type most resembling the session in the laboratory | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Among a predetermined list of gambling location type (e.g. bar/restaurant, casino, etc.), participant choose which the gambling session in the laboratory resembled the most.
Perceived realism - Session in the laboratory VS gambling on EGMs in a bar/restaurant | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Level on resemblance between a gambling session on EGMs in a bar/restaurant and the gambling session in the laboratory. Evaluated with a 7-points Likert scale (1 = "Almost 100 % different" to 7 = "Almost 100 % the same").
Perceived realism - Similarities between session in the laboratory VS gambling on EGMs in a bar/restaurant | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Things that were the same or very alike when comparing a gambling session on EGMs in a bar/restaurant and the gambling session in the laboratory. Participant lists all resemblances that come to their mind.
Perceived realism - Differences between session in the laboratory VS gambling on EGMs in a bar/restaurant | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Things that were not the same or very not alike when comparing a gambling session on EGMs in a bar/restaurant and the gambling session in the laboratory. Participant lists all differences that come to their mind.
Perceived realism - What could be done to heighten realism of the session in the laboratory | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Things or aspects of the study that be changed in order for the gambling session in the laboratory to be more alike a real gambling session on EGMs in a bar/restaurant. Participant lists all that come to their mind.
Perceived realism - Effect of using one own money on realism | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Effect of gambling one own money in this study on the level of realism. Evaluated with a 7-points Likert scale (1 = "It lessened the realism a lot" to 7 = " It heighten the realism a lot ").
Perceived realism - Effect of using one own money on realism (free) | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Effect of gambling one own money in this study on the level of realism. Participant freely explain their perception of said effect.
Perceived correspondence between habitual gambling behaviour and gambling behaviour during the session in the laboratory | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Participant's perception of how much their gambling behaviour during their gambling session in the laboratory was representative (i.e. how much it was the same) of their gambling behaviour on EGMs in the past 12 months. Evaluated with a 7-points Likert scale (1 = "Almost 100 % different" to 7 = "Almost 100 % the same").
Perceived correspondence between habitual gambling behaviour and gambling behaviour during the session in the laboratory (free) | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Participant's perception of how much their gambling behaviour during their gambling session in the laboratory was representative (i.e. how much it was the same) of their gambling behaviour on EGMs in the past 12 months. Participant freely explain their perception.
Protocol credibility | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Participant's level of certitude they were betting their own money and that they could loose money for real during the study. Evaluated with a 7-points Likert scale (1 = "Almost 100 % certain they were going to get their money back at the end of the study" to 7 = "Almost 100 % certain winnings and losses were real").
Protocol credibility (free) | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Participant comment freely on their level of certitude that they were betting their own money and that they could loose money for real during the study.
Recruitment potential - Volunteers | Assessed after recruitment for the study is ended (80 participants recruited) or 1 year after recruitment for the study has begun, whichever came first.
  Number of people that answered the recruitment ad and wanted to either participate or get more information on the study.
Recruitment potential - Recruited | Assessed after recruitment for the study is ended (80 participants recruited) or 1 year after recruitment for the study has begun, whichever came first.
  Number of people that qualified and agreed to participate in the study.
Recruitment potential - Rejected | Assessed after recruitment for the study is ended (80 participants recruited) or 1 year after recruitment for the study has begun, whichever came first.
  Number of people that volunteered to participate but didn't qualify according to the inclusion/exclusion criteria.
Recruitment potential - Refusal | Assessed after recruitment for the study is ended (80 participants recruited) or 1 year after recruitment for the study has begun, whichever came first.
  Number of people that qualified for participation in the study but refused to do so after hearing the details of it.
Attrition | Assessed after recruitment for the study is ended (80 participants recruited) or 1 year after recruitment for the study has begun, whichever came first.
  Number of people that qualified and agreed to participate in the study but desisted during their participation.

OTHER OUTCOMES:
Prevention pop-up messages recall - Free recall (Y/N) | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Participant is asked if they saw any prevention pop-up messages during their gambling session in the laboratory. This is a Yes/No question.
Prevention pop-up messages recall - Free recall (number) | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  If participant declared they saw prevention pop-up messages during their gambling session in the laboratory, they are asked how many there were. The same message presented twice count as "2".
Prevention pop-up messages recall - Free recall (content) | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  If participant declared they saw prevention pop-up messages during their gambling session in the laboratory, they are asked to freely describe them (i.e. content, graphical appearance, etc.).
Prevention pop-up messages recall - Cued recall (Y/N) | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  Participant is presented with a list of prevention pop-up messages that could have been shown during the study. For each of them, they are asked to identify if they saw it or no.
Prevention pop-up messages recall - Cued recall (number) | Assessed at the end gambling session in the laboratory (Post-experiment phase). Session's length is decided by participant (but limited to 2 hours maximum).
  If participant declared they saw prevention pop-up messages during their gambling session in the laboratory, they are asked how many there were. The same message presented twice count as "2". This is different from Outcome 39 because, participant might recognize a message they had forgotten about or a message they saw but didn't considered it a "prevention message".

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Galipeau, Principal Investigator — Laval University
Locations (1):
- Centre québécois d'excellence pour la prévention et le traitement du jeu, Québec, Canada

IPD SHARING:
Plan to Share IPD: No
The ethics committee doesn't allow for unrestricted sharing of IPD. However, we will try our best to answer any questions related to IPD within the boundaries set by the ethics committee.

REFERENCES:
- [Background] Dillard JP, Shen L. On the nature of reactance and its role in persuasive health communication. Communication monographs. 2005; 72(2): 144-168.
- [Background] Ferris J, Wynne H. The Canadian Problem Gambling Index: Final Report. 2001. https://www.greo.ca/Modules/EvidenceCentre/files/Ferris%20et%20al(2001)The_Canadian_Problem_Gambling_Index.pdf
- [Background] Delfabbro P, King DL, Browne M, Dowling NA. Do EGMs have a Stronger Association with Problem Gambling than Racing and Casino Table Games? Evidence from a Decade of Australian Prevalence Studies. J Gambl Stud. 2020 Jun;36(2):499-511. doi: 10.1007/s10899-020-09950-5. PMID 32306234
- [Background] Bjorseth B, Simensen JO, Bjornethun A, Griffiths MD, Erevik EK, Leino T, Pallesen S. The Effects of Responsible Gambling Pop-Up Messages on Gambling Behaviors and Cognitions: A Systematic Review and Meta-Analysis. Front Psychiatry. 2021 Jan 25;11:601800. doi: 10.3389/fpsyt.2020.601800. eCollection 2020. PMID 33569015
- [Background] Ginley MK, Whelan JP, Pfund RA, Peter SC, Meyers AW. Warning messages for electronic gambling machines: evidence for regulatory policies. Addiction Research & Theory. 2017; 25(6): 495-504. doi: 10.1080/16066359.2017.1321740
- [Background] Livingstone C, Rintoul A, Francis L. What is the evidence for harm minimisation measures in gambling venues? Evidence Base: A Journal of Evidence Reviews in Key Policy Areas. 2014; (2), 1-24. https://search.informit.org/doi/10.3316/informit.
- [Background] Williams RJ, West BL, Simpson RI. Prevention of problem gambling: A comprehensive review of the evidence and identified best practices. 2012. https://opus.uleth.ca/bitstream/handle/10133/3121/2012-PREVENTION-OPGRC.pdf?sequence=3&isAllowed=y
- [Background] MacLaren VV. Video Lottery is the Most Harmful Form of Gambling in Canada. J Gambl Stud. 2016 Jun;32(2):459-85. doi: 10.1007/s10899-015-9560-z. PMID 26233645
- [Background] Papineau E, Lacroix G, Sevigny S, Biron JF, Corneau-Tremblay N, Lemétayer F. Assessing the differential impacts of online, mixed, and offline gambling. International Gambling Studies. 2018; 18(1): 69-91. doi: 10.1080/14459795.2017.1378362
- [Background] Billieux J, Van der Linden M, Khazaal Y, Zullino D, Clark L. Trait gambling cognitions predict near-miss experiences and persistence in laboratory slot machine gambling. Br J Psychol. 2012 Aug;103(3):412-27. doi: 10.1111/j.2044-8295.2011.02083.x. Epub 2011 Oct 24. PMID 22804705
- [Background] Blaszczynski A, Cowley E, Anthony C, Hinsley K. Breaks in Play: Do They Achieve Intended Aims? J Gambl Stud. 2016 Jun;32(2):789-800. doi: 10.1007/s10899-015-9565-7. PMID 26275785
- [Background] Floyd K, Whelan JP, Meyers AW. Use of warning messages to modify gambling beliefs and behavior in a laboratory investigation. Psychol Addict Behav. 2006 Mar;20(1):69-74. doi: 10.1037/0893-164X.20.1.69. PMID 16536667
- [Background] Harris A, Parke A. The Interaction of Gambling Outcome and Gambling Harm-Minimisation Strategies for Electronic Gambling: the Efficacy of Computer Generated Self-Appraisal Messaging. International Journal of Mental Health and Addiction. 2016; 14(4): 597-617. doi: 10.1007/s11469-015-9581-y
- [Background] Cloutier M, Ladouceur R, Sevigny S. Responsible gambling tools: pop-up messages and pauses on video lottery terminals. J Psychol. 2006 Sep;140(5):434-8. doi: 10.3200/JRLP.140.5.434-438. PMID 17066750
- [Background] Kim HS, Wohl MJ, Stewart MJ, Sztainert T, Gainsbury SM. Limit your time, gamble responsibly: Setting a time limit (via pop-up message) on an electronic gaming machine reduces time on device. International Gambling Studies. 2014; 14(2): 266-278. doi: 10.1080/14459795.2014.910244
- [Background] Ladouceur R, Sévigny S. Interactive messages on video lottery terminals and persistence in gambling. Gambling Research. 2003; 15(1): 44-49.
- [Background] Brandt AE, Sztykiel H, Pietras CJ. Laboratory simulated gambling: risk varies across participant-stake procedure. J Gen Psychol. 2013 Apr-Jun;140(2):130-43. doi: 10.1080/00221309.2013.776509. PMID 24837532
- [Background] Anderson G, Brown RI. Real and laboratory gambling, sensation-seeking and arousal. Br J Psychol. 1984 Aug;75 ( Pt 3):401-10. doi: 10.1111/j.2044-8295.1984.tb01910.x. PMID 6487928
- [Background] Ladouceur R, Gaboury A, Bujold A, Lachance N, Tremblay S. Ecological validity of laboratory studies of videopoker gaming. J Gambl Stud. 1991 Jun;7(2):109-16. doi: 10.1007/BF01014526. PMID 24242983
- [Background] Weatherly JN, Brandt AE. Participants' sensitivity to percentage payback and credit value when playing a slot-machine simulation. Behavior and Social Issues. 2004; 13(1): 33-51.doi: 10.5210/bsi.v13i1.34
- [Background] Weatherly JN, McDougall CL, Gillis AA. A bird in hand: discouraging gambling on a slot machine simulation. J Psychol. 2006 Jul;140(4):347-61. doi: 10.3200/JRLP.140.4.347-361. PMID 16967741
- [Background] Weatherly JN, Meier E. Studying gambling experimentally: The value of money. Analysis of Gambling Behavior. 2007; 1(2): article 5. https://repository.stcloudstate.edu/agb/vol1/iss2/5